CLINICAL TRIAL: NCT04033887
Title: Evaluation Study of Rapid Diagnostic Tests (RDTs) Detecting Antibodies Against Hepatitis C Virus
Brief Title: Evaluation Study of RDTs Detecting Antibodies Against HCV
Status: Completed | Type: Observational
Sponsor: Foundation for Innovative New Diagnostics, Switzerland (Other)
Collaborators: Institute of Tropical Medicine, Belgium (Other); Nigerian Institute of Medical Research (Other Government); Richard Lugar Centre for Public Health Research, Georgia (Unknown)
Responsible Party: Sponsor
Other Study IDs: 8162-2/1
Record Dates: First submitted 2019-03-18; First posted 2019-07-26 (Actual); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Hepatitis C
Keywords: Diagnosis; HIV coinfection; Rapid diagnostic test
MeSH Terms: conditions — Hepatitis C; Disease; HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HCV-only infected: Archived frozen plasma samples from individuals that were characterised to be HCV-antibody positive or HCV-antibody negative ("HCV-only infected"). These samples are characterised for their HIV status (negative).
  Interventions: Diagnostic Test: 13 Rapid Diagnostic Tests and reference tests
- HCV/HIV co-infected: Archived frozen plasma samples from HCV-positive or HCV-negative individuals who are HIV infected ("HCV/HIV co-infected").
  Interventions: Diagnostic Test: 13 Rapid Diagnostic Tests and reference tests

INTERVENTIONS:
Diagnostic Test: 13 Rapid Diagnostic Tests and reference tests — Rapid diagnostic tests:
  1. HCV antibody test (under development); bioLytical Laboratories
  2. DPP® HCV (under development); Chembio Diagnostic Systems
  3. HCV-Ab Rapid Test; Beijing Wantai Biological Pharmacy Enterprise
  4. Rapid Anti-HCV Test; InTec
  5. First Response HCV Card Test; Premire Medical Corporation
  6. Signal HCV Ver 3.0; Arkray healthcare
  7. TRI DOT HCV; J. Mitra & Co
  8. Triplex HIV, HCV, HBsAg; Biosynex SA
  9. Standard Q HCV Ab; SD Biosensor
  10. HCV Hepatitis Virus Antibody Test; Artron Laboratories
  11. SD Bioline HCV; Abbott Diagnostics
  12. OraQuick HCV; OraSure
  13. Care Start HCV Rapid Test (under development); Access Bio
  Reference tests:
  Enzyme Immunoassays (EIAs): Murex Anti-HCV EIA version 4.0; Fujirebio Innotest HCV Ab IV
  Line Immunoassay (LIA): MP Diagnostics HCV blot 3.0

SUMMARY:
The study aims to evaluate 13 different HCV RDTs (10 on-market, 3 under development) for their diagnostic performance and operational characteristics in archived EDTA plasma samples, originating from patients from different geographical regions (Nigeria, Georgia, Cambodia, Belgium) and with or without HIV co-infection.

DETAILED DESCRIPTION:
Background and rationale:

Screening of past exposure to Hepatitis C Virus (HCV) infection is done by detection of HCV specific antibodies. In Low and Middle Income Countries (LMICs), where equipped laboratories and trained staff are limited, Rapid Diagnostic Tests (RDTs) are widely used for HCV screening. Although many RDTs are available on the market, only some of them received CE-IVD marking and only two have been validated by WHO Pre-Qualification (PQ). More quality-assured tests are needed to establish effective screening programmes in LMICs.

Furthermore, an important research gap is the lack of studies on the impact of HIV positivity on RDT performance, as it is estimated that 2-15% of people living with HIV are co-infected with HCV.

The evaluation of RDT performance on clinical samples collected in different geographic regions as well as from HIV co-infected individuals, would allow to identify tests with a performance meeting or having the potential to meet WHO quality standards.

Concept:

This is a multicenter laboratory evaluation study using archived, frozen plasma samples.

Sensitivity and specificity of RDTs will be measured against a composite reference standard that consists of two WHO prequalified Enzyme Immunoassays (EIAs) (Murex Anti-HCV EIA version 4.0, Fujirebio Innotest HCV Ab IV) and a Line Immunoassay (LIA) (MP Diagnostics HCV blot 3.0). Samples are assigned as anti-HCV negative or anti-HCV positive based on the results of all three assays.

RDT results will be read by three independent readers to evaluate inter-reader variability (differences in visual interpretation, i.e. presence or absence of test and control line).

For each RDT, two independently produced lots will be tested for each sample to assess lot-to-lot variability (differences in RDT result for the same sample). Furthermore, rate of invalid runs will be assessed and a technical appraisal is completed for each RDT.

Primary objective:

1.1 Evaluation of sensitivity and specificity of anti-HCV RDTs in archived plasma samples, collected from HCV-infected and HCV-uninfected individuals not co-infected with HIV, measured against the composite reference standard composed of two Enzyme Immunoassays (EIAs) and a Line Immunoassay (LIA).

1.2 Evaluation of sensitivity and specificity of anti-HCV RDTs in archived plasma samples, collected from HCV-infected and HCV-uninfected individuals who are all co-infected with HIV, measured against the composite reference standard composed of two EIAs and a LIA.

Secondary objectives:

2.1 Evaluation of sensitivity and specificity of anti-HCV RDTs in archived plasma samples, collected from HCV-infected and HCV-uninfected individuals, both co-infected and not with HIV, measured against the composite reference standard composed of two EIAs and a LIA.

2.2 Evaluation of operational characteristics of anti-HCV RDTs: inter-reader variability; lot-to-lot variability; rate of invalid runs 2.3 Technical appraisal of each RDT product per manufacturer

ELIGIBILITY:
Inclusion Criteria of archived samples:

* Non-hemolytic plasma samples with EDTA used as anticoagulant
* Sample were frozen at -20°C or lower on the day of processing and stored at -20°C or lower until they are used in this study
* Samples pre-characterized for, HCV, HIV serology status using assays routinely used at the sites and approved for diagnostic use by a local health authority. If available, samples should also be characterized for HBV status.
* Samples taken from subjects aged ≥18 years
* Availability of informed consent to use the sample in future research

Exclusion Criteria:

- Samples not stored correctly

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Samples tested in Belgium originate from Cambodia (80%) and Belgium (20%). Cambodian samples are leftovers from samples collected during a cross-sectional study of hepatitis C among people living with HIV (De Weggheleire, A. 2017); samples in Belgium were collected and archived during routine patient care visits to the HIV clinic.
  Samples in Nigeria originate from routine diagnostic activities at NIMR as well as the AIDS Prevention Initiative Nigeria (APIN) PEPFAR Program Sample/Data Bank setup at NIMR and the Lagos University Teaching Hospital.
  Samples tested in Georgia are leftover samples from a previous FIND HCV study (Reipold, E.I., 2019), as well as archived routine diagnostic samples from the site.
  Percent sample distribution per site:
  Belgium: 38% Nigeria: 41% Georgia: 21%
Sampling Method: Probability Sample
Enrollment: 1710 (Actual)
Dates: Start 2018-09-21 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-03-15 (Actual)

PRIMARY OUTCOMES:
Point estimates of sensitivity and specificity, with 95% confidence intervals, of RDTs for the detection of anti-HCV antibodies in individuals not co-infected with HIV. | 6 months
  Point estimates of sensitivity and specificity, with 95% confidence Intervals based on Wilson's score method, will be computed for all samples HCV+ve/HIV-ve and HCV-ve/HIV-ve; the calculation was performed for all RDT manufacturers and individually for each lot. The estimates were calculated on the overall sample population.
Point estimates of sensitivity and specificity, with 95% confidence intervals, of RDTs for the detection of anti-HCV antibodies in HIV co-infected individuals. | 6 months
  Point estimates of sensitivity and specificity, with 95% confidence Intervals based on Wilson's score method, were computed for all samples HCV+ve/HIV+ve and HCV-ve/HIV+ve; the calculation was performed for all RDT manufacturers and individually for each lot. The estimates were calculated on the overall sample population.

SECONDARY OUTCOMES:
Point estimates of sensitivity and specificity, with 95% confidence intervals, of RDTs for the detection of anti-HCV antibodies in the overall sample population. | 6 months
  Point estimates of sensitivity and specificity, with 95% confidence intervals based on Wilson's score method, were computed for all samples: HCV+ve/HIV-ve, HCV-ve/HIV-ve, HCV+ve/ HIV+ve and HCV-ve/HIV+ve; the was performed for all RDT manufacturers and individually for each lot. The estimates were calculated on the overall sample population.
Operational characteristics | 6 months
  Inter-reader variability: Fleiss Kappa Coefficient (κ) of inter-reader variability per RDT; manufacturer lot Lot-to-lot variability: coefficient of lot-to-lot variability (percentage agreement) per RDT manufacturer Rate of invalid runs: Percent of invalid runs per manufacturer lot
Technical appraisal rating on kit instructions, packaging, labelling and test conduct, on a Likert scale | 6 months
  Averages of likert-scale scores will be calculated and serve to understand the user-friendliness of the RDT; there is no expected outcome, the scale rating is used to collect consistent feedback from users; scale scores are as follows: 1=poor, 2=needs improvement, 3=satisfactory, 4=good, 5=excellent

CONTACTS AND LOCATIONS:
Overall Officials: Ranga Sampath, PhD, Study Director — Foundation for Innovative New Diagnostics, Geneva, Switzerland; Rosemary Audu, PhD, Principal Investigator — Nigerian Institute of Medical Research, Lagos, Nigeria; Katrien Fransen, PhD, Principal Investigator — Institute of Tropical Medicine, Antwerp, Belgium; Maia Alkhazashvili, Masters, Principal Investigator — NCDC Lugar Centre, Tbilisi, Georgia
Locations (3):
- Institute of Tropical Medicine, Antwerp, Belgium
- National Center for Disease Control & Public Health/Lugar Center, Tbilisi, Georgia
- Nigerian Institute of Medical Research, Lagos, Nigeria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] De Weggheleire A, An S, De Baetselier I, Soeung P, Keath H, So V, Ros S, Teav S, Smekens B, Buyze J, Florence E, van Griensven J, Thai S, Francque S, Lynen L. A cross-sectional study of hepatitis C among people living with HIV in Cambodia: Prevalence, risk factors, and potential for targeted screening. PLoS One. 2017 Aug 23;12(8):e0183530. doi: 10.1371/journal.pone.0183530. eCollection 2017. PMID 28832660
- [Background] Reipold, E.I., Evaluation of the diagnostic performance of the Xpert® Fingerstick HCV Viral Load (VL) Assay. Manuscript in preparation 2019
- [Derived] Vetter BN, Reipold EI, Ongarello S, Audu R, Ige FA, Alkhazashvili M, Chitadze N, Vanroye F, De Weggheleire A, An S, Fransen K. Sensitivity and Specificity of Rapid Diagnostic Tests for Hepatitis C Virus With or Without HIV Coinfection: A Multicentre Laboratory Evaluation Study. J Infect Dis. 2022 Aug 26;226(3):420-430. doi: 10.1093/infdis/jiaa389. PMID 32614451